CLINICAL TRIAL: NCT00205686
Title: DHEA+Exercise-Effect on Sarcopenia and Osteopenia of Aging
Brief Title: Effects of DHEA and Exercise in the Elderly
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: K23RR016191 (NIH); K23RR016191 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2006-01-06 (Estimated); Status verified 2005-09

CONDITIONS: Healthy Volunteers
Keywords: Aging, dhea, bone density, muscle mass, insulin action
MeSH Terms: interventions — Dehydroepiandrosterone; Exercise

INTERVENTIONS:
Drug: DHEA
Behavioral: exercise

SUMMARY:
DHEA or dehydroepiandrosterone is a naturally occurring hormone secreted by tghe adrenal galnds. The secretion of HDEA declines with aging. DHEA is considered a food supplement and it is not regulated by the FDA. The purpose of this research is to evaluate ceratin of the biological effects of a reaplcement dose of DHEA. As you get older, DHEA levels are lower than you were younger. The replamcent dose is the dose of DHEA that will raise DHEA levesl to the levels found in young people. Anotehr purpose is to determine whether DHEA enhances the adaptations to an exercise training program.

DETAILED DESCRIPTION:
DHEA declines dramatically with age. Low DHEA levels have been found to correlate with sarcopenia and osteopenia. It is, therefore, postulated that many physiologic changes of aging are secondary to the decline in DHEA. Thus, the objective of the proposed research is to evaluate the effect of DHEA replacement on age-related changes in body composition, muscle function and metabolism, and bone mass in healthy older adults. The specific aims are to evaluate the effects of DHEA replacement (50 mg/d) alone, or in combination with resistance exercise training on: a) lean body mass, intraabdominal fat and thigh muscle volume, and muscle protein synthesis rate b) bone mineral density (BMD) of the total body, lumbar spine, and hip and biochemical markers of bone turnover and c) insulin sensitivity. It is hypothesized that DHEA administration will have additive or synergistic effects with exercise. Healthy but sedentary subjects , aged 65-78 years old, will be randomized to receive either DHEA, 50 mg/d, or placebo and to participate in either supervised or home exercise training programs. The supervised exercise program will consist of resistance training designed to increase muscle mass, strength, and bone mass, and decrease fat mass. The goal of this research is to provide information on the potential role of DHEA replacement therapy in maintaining the physical health and functional capacity of older people

ELIGIBILITY:
Inclusion Criteria:

* 65 to 78 years old men and women

Exclusion Criteria:

* hormone therapy, history of hormone-dependent neoplasia, PSA above 2.6 ng/mL, or active serious illness, contraindications to exercise, dementia

Ages: 65 Years to 78 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 64
Dates: Start 2001-04; Study Completion 2005-09

PRIMARY OUTCOMES:
thigh muscle mass, muscle strength, intadominal fat, bone mineral density, markers of bone turnover, insulin sensitivity,

SECONDARY OUTCOMES:
quality of life, vascular reactivity, levels of hormones

CONTACTS AND LOCATIONS:
Overall Officials: Dennis T Villareal, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Villareal DT, Holloszy JO, Kohrt WM. Effects of DHEA replacement on bone mineral density and body composition in elderly women and men. Clin Endocrinol (Oxf). 2000 Nov;53(5):561-8. doi: 10.1046/j.1365-2265.2000.01131.x. PMID 11106916
- [Background] Villareal DT. Effects of dehydroepiandrosterone on bone mineral density: what implications for therapy? Treat Endocrinol. 2002;1(6):349-57. doi: 10.2165/00024677-200201060-00001. PMID 15832488
- [Result] Villareal DT, Holloszy JO. Effect of DHEA on abdominal fat and insulin action in elderly women and men: a randomized controlled trial. JAMA. 2004 Nov 10;292(18):2243-8. doi: 10.1001/jama.292.18.2243. PMID 15536111